CLINICAL TRIAL: NCT01582399
Title: A Phase 1 Single-Dose, Parallel Group, Randomized, Open-Label Study to Determine the Absolute Bioavailability of ASKP1240 After Intravenous and Subcutaneous Administration in Healthy Subjects
Brief Title: Bioavailability of ASKP1240 in Healthy Subjects After Intravenous and Subcutaneous Administration of ASKP1240
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Collaborators: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 7163-CL-0106
Record Dates: First submitted 2012-04-19; First posted 2012-04-20 (Estimated); Last update posted 2012-12-10 (Estimated); Status verified 2012-12

CONDITIONS: Pharmacokinetics of ASKP1240; Pharmacodynamics of ASKP1240; Healthy Volunteers
Keywords: Healthy Volunteers; CD40 receptor occupancy; Co-stimulation blockade; CD40 antigen; Anti-CD40; ASKP1240
MeSH Terms: interventions — bleselumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A: ASKP1240 intravenous (IV) infusion (Experimental)
  Interventions: Drug: ASKP1240
- Arm B: ASKP1240 subcutaneous (SC) (Experimental)
  Interventions: Drug: ASKP1240

INTERVENTIONS:
Drug: ASKP1240 — intravenous(IV) infusion and subcutaneous (SC)

SUMMARY:
The objective of this study is to assess levels of ASKP1240 in the blood after a single dose given intravenously (IV) or as a subcutaneous (SC) injection. The study will determine how the drug behaves inside the body and how it is eliminated from the body by looking at the pharmacokinetics of ASP1240.

In addition, the study will determine the effects of ASKP1240 on the body by looking at its pharmacodynamics (PD) and at the safety and tolerability of ASKP1240 when given by IV or as SC injection.

ELIGIBILITY:
Inclusion Criteria:

* The subject weighs at least 50 kg, and has a body mass index (BMI) of 18 to 32 kg/m2, inclusive
* The female subject must be a) at least two years post-menopausal (defined as at least 2 years without menses) at Screening and a confirmatory follicle stimulating hormone (FSH) level of >40 U/L at Screening) or b) surgically sterile (with documentation provided by a healthcare professional) and not pregnant or lactating at Screening and Day -1. c) If child bearing potential, the subject will be required to use adequate contraception consisting of two forms of birth control (one of which must be a barrier method) until the end of the study or for 90 days after final study drug administration, whichever is longer
* The male subject agrees to sexual abstinence, is surgically sterile (with documentation provided by a healthcare professional), or is using a medically acceptable method (e.g. spermicide and diaphragm, or spermicide and condom) to prevent pregnancy and agrees to continue using this method until the end of study
* Male subject agrees to no sperm donation until the end of the study or for 90 days after the conclusion of study drug administration, whichever is longer

Exclusion Criteria:

* The subject has a history or evidence of any clinically significant (as determined by the Investigator) cardiovascular, endocrine, ophthalmologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary (including asthma or emphysema), neurologic, dermatologic, psychiatric, renal, and/or other major disease or malignancy (excluding non-melanoma skin cancer)
* The subject has a history of severe allergic or anaphylactic reactions
* The subject has a history of consuming more than 14 units of alcoholic beverages (one unit is 12 ounces of beer, 4 ounces of wine or 1 ounce of spirits) per week on average within 6 months prior to Screening or has a history of alcoholism or drug/chemical/substance abuse within past 2 years prior to Screening or the subject tests positive at Screening or Day -1 for alcohol or drugs of abuse (amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, and opiates)
* The subject has/had a symptomatic, viral, bacterial or fungal (non-cutaneous) infection within 1 week prior to clinic check in on Day -1
* The subject has a history of thromboembolic or vascular disease especially deep vein thrombosis or pulmonary embolism
* The subject has used any tobacco-containing products, nicotine or nicotine-containing products in the past 6 months prior to Screening
* The subject has a supine mean systolic blood pressure < 90 or > 160 mmHg and a mean diastolic blood pressure < 50 or > 90 mmHg, or mean heart rate > 100 beats per minute (bpm), either at Screening or Day -1 (measurements taken in triplicate after subject has been resting in a supine position for a minimum of 5 minutes)
* The subject is known to be positive for human immunodeficiency virus (HIV) antibody
* The subject has a positive test for hepatitis C virus (HCV) antibody, hepatitis B surface antigen (HBsAg), or hepatitis B core antibody at Screening
* The subject has the following at Screening or Day -1:

  1. White blood cell count (WBC) is < 3.5 (109/L) or > upper limit of normal
  2. Absolute neutrophil count (ANC) is < 1.5 (109/L) or > upper limit of normal
  3. Platelet count (PLT) is outside the normal limit
  4. Serum creatinine, total bilirubin, alanine aminotransferase (ALT), or aspartate aminotransferase (AST) are > upper limit of normal
  5. Creatine phosphokinase (CPK) is > 2x times upper limit of normal
  6. International normalized ratio (INR) is > upper limit of normal
  7. Remaining laboratory tests are outside the normal limits and considered by the investigator to be clinically significant with regard to the remaining per-protocol laboratory tests
* The subject has received any vaccine within 60 days prior to Day -1
* The subject has received any systemic immunosuppressant agent (e.g., methotrexate) within 6 months prior to Day -1
* The subject has received any systemic steroid within 2 months prior to Day -1
* The subject has received any antibody or therapeutic biologic product within 6 months prior to Day -1
* The subject has used prescription or non-prescription medications (excluding acetaminophen [up to 2 g/day maximum], stable hormone replacement therapy [HRT], and/or nasal steroids/steroid inhaler), or complementary and alternative medicines (CAM) within 14 days or 5 half lives (whichever is longer) prior to Day -1
* The subject has a positive TB skin test, Quantiferon Gold test or T-SPOT test® at Screening
* The subject has participated in a previous ASKP1240 study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2012-02; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic profile: AUClast, AUCinf, and F | Day 15 to Day 90, ± 3 days
  Area under the serum concentration- time curve from time 0 up to the last quantifiable concentration (AUClast), Area under the serum concentration- time curve from time 0 extrapolated to infinity (AUCinf), and Absolute bioavailability (F)

SECONDARY OUTCOMES:
Pharmacodynamic profile: CD40 receptor occupancy over time | Day 15 to Day 90, ± 3 days
  Cell surface antigen, target of ASKP1240 (CD40), as measured on CD20+ B lymphocytes
Pharmacodynamic profile: Total lymphocyte count and peripheral lymphocyte subset quantification | Day 15 to Day 90, ± 3 days
  Total lymphocyte count = product of the white blood count (WBC) and percent lymphocytes [from differential]
Pharmacokinetics profile: Cmax, Tmax, t1/2, Vz, and CLtot | Day 15 to Day 90, ± 3 days
  Maximum concentration (Cmax),Time to attain Cmax (Tmax), Apparent terminal elimination of half-life (t1/2), Apparent volume of distribution ( Vz), and Total body clearance (CLtot)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development
Locations (1):
- Parexel, Baltimore, Maryland, United States